CLINICAL TRIAL: NCT00931138
Title: Treatment of AML in Adults 50 to 70 Years, Study of Two Anthracyclines and the Interest of Maintenance Treatment With Interleukin 26- ALFA 9801
Brief Title: Treatment of Acute Myeloid Leukemia (AML) in Adults 50 to 70 Years, Study of Two Anthracyclines and the Interest of Maintenance Treatment With Interleukin 2
Acronym: ALFA 9801
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acute Leukemia French Association (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Pr Sylvie Castaigne - Pricipal Investigator, CHV A. MIGNOT
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFA 9801
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 1999-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia in adults; Newly-diagnosed untreated AML; Patient aged 50 to 70 years
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm1 = Aracytine + Daunorubicin (Active Comparator): Aracytine : 200 mg/m2 d1-d7 Daunorubicin : 80 mg/m2 d1-d3
  Interventions: Drug: chemotherapy (Aracytine + Daunorubicin)
- Arm 3 = Aracytine And Idarubicin (Active Comparator): Aracytine : 200 mg/m2 d1-d7 Idarubicin : 12 mg/m2 d1-d4
  Interventions: Drug: chemotherapy (Aracytine + Daunorubicin)
- Arm 2 = Aracytine And Idarubicin (Active Comparator): Aracytine : 200 mg/m2 d1-d7 Idarubicin :12 mg/m2 d1-d3
  Interventions: Drug: chemotherapy (Aracytine + Daunorubicin)

INTERVENTIONS:
Drug: chemotherapy (Aracytine + Daunorubicin) — Aracytine : 200 mg/m2 d1-d7 Daunorubicin : 80 mg/m2 d1-d3
  Arms: Arm1 = Aracytine + Daunorubicin
Drug: chemotherapy (Aracytine + Daunorubicin) — Aracytine : 200 mg/m2 d1-d7 Idarubicin :12 mg/m2 d1-d3
  Arms: Arm 2 = Aracytine And Idarubicin
Drug: chemotherapy (Aracytine + Daunorubicin) — Aracytine : 200 mg/m2 d1-d7 Idarubicin : 12 mg/m2 d1-d4
  Arms: Arm 3 = Aracytine And Idarubicin

SUMMARY:
Randomized comparison of standard induction treatment with daunorubicin for 3 days and Idarubicin for 3 or 4 days in adult AML patients between 50 and 70 years. Study of maintenance treatment with IL2

DETAILED DESCRIPTION:
Patients from 50 to 70 years with de novo AML were randomized to receive ARAC 200 mg / m² / d IV x 7 d with either DNR 80 mg/m²/dx3d (arm 1) or IDA 12 mg / m²/d x 3 d (arm 2) or 4 d (arm 3). The pts received a failing course of remedial Mitoxantrone involving x 2 and j ARAC 1g / m 2 x / d x 4 days The pts in CR then received 2 courses of consolidation with, according to initial randomization either DNR 80 mg / m² IDA 12 mg / sqm x 1 d (1st treatment) or 2 d (2nd treatment) and ARAC 1 gsm 2/jx x 4 days The pts in CR were then randomized persistent IL2 (5 million IU / m² x 5 d / month in SC for 12 months) or no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 50 to 70 years
* AML de Novo
* No prior therapy for AML
* Absence of severe infection (WHO grade greater than 2), independent of the AML
* Cardiac function determined by radionucleotide or echography within normal limits.
* total bilirubin less than or equal 2N and Serum creatinin less than or equal 2N
* ECOG performance status 0 to 3
* Signed informed consent.

Exclusion Criteria:

* M3-AML
* history of neoplasia treated by radiotherapy or chemotherapy
* Myelodysplasia diagnosed more than 6 months before the diagnosis of AML
* Prior treatment for AML
* Uncontrolled infection
* Other active malignancy
* Patient unable to undergo regular surveillance

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 1999-12; Study Completion 2006-12

PRIMARY OUTCOMES:
To compare idarubicin versus daunorubicin: the duration of the event-free survival (EFS) to compare IL2 versus abstention : the relapse rate assessed during the first year following the start of maintenance treatment with interleukin

SECONDARY OUTCOMES:
Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CH, Caen
  - Hopital Percy, Clamart
  - CHU, Créteil
  - CH, Lens
  - CHU, Lille
  - CH, Limoges
  - Hopital Edouard Herriot, Lyon
  - St Antoine Hospital, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Saint-Louis, Paris
  - CH, Roubaix
  - CHU, Rouen
  - CNLCC, Saint-Cloud
  - CH, Valenciennes
  - CH, Versailles
  - IGR, Villejuif

REFERENCES:
- [Derived] Sarkozy C, Gardin C, Gachard N, Merabet F, Turlure P, Malfuson JV, Pautas C, Micol JB, Thomas X, Quesnel B, Celli-Lebras K, Preudhomme C, Terre C, Fenaux P, Chevret S, Castaigne S, Dombret H. Outcome of older patients with acute myeloid leukemia in first relapse. Am J Hematol. 2013 Sep;88(9):758-64. doi: 10.1002/ajh.23498. Epub 2013 Aug 7. PMID 23749683
- [Derived] Gardin C, Chevret S, Pautas C, Turlure P, Raffoux E, Thomas X, Quesnel B, de Revel T, de Botton S, Gachard N, Renneville A, Boissel N, Preudhomme C, Terre C, Fenaux P, Bordessoule D, Celli-Lebras K, Castaigne S, Dombret H. Superior long-term outcome with idarubicin compared with high-dose daunorubicin in patients with acute myeloid leukemia age 50 years and older. J Clin Oncol. 2013 Jan 20;31(3):321-7. doi: 10.1200/JCO.2011.40.3642. Epub 2012 Dec 17. PMID 23248249
- [Derived] Itzykson R, Gardin C, Pautas C, Thomas X, Turlure P, Raffoux E, Terre C, Fenaux P, Castaigne S, Dombret H, Boissel N; Acute Leukemia French Association (ALFA). Impact of post-remission therapy in patients aged 65-70 years with de novo acute myeloid leukemia: a comparison of two concomitant randomized ALFA trials with overlapping age inclusion criteria. Haematologica. 2011 Jun;96(6):837-44. doi: 10.3324/haematol.2010.036921. Epub 2011 Apr 1. PMID 21459791
- [Derived] Boissel N, Nibourel O, Renneville A, Gardin C, Reman O, Contentin N, Bordessoule D, Pautas C, de Revel T, Quesnel B, Huchette P, Philippe N, Geffroy S, Terre C, Thomas X, Castaigne S, Dombret H, Preudhomme C. Prognostic impact of isocitrate dehydrogenase enzyme isoforms 1 and 2 mutations in acute myeloid leukemia: a study by the Acute Leukemia French Association group. J Clin Oncol. 2010 Aug 10;28(23):3717-23. doi: 10.1200/JCO.2010.28.2285. Epub 2010 Jul 12. PMID 20625116